CLINICAL TRIAL: NCT02132988
Title: An Open Labeled Phase II Trial of Active Immunotherapy With Globo H-KLH (OPT-822/821) in Women Who Have Non-Progressive Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Trial of Active Immunotherapy With Globo H-KLH (OPT-822/821) in Women Who Have Non-Progressive Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: OBI Pharma, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMH-OPT822-OC001
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPT-822/OPT-821 (Experimental)
  Interventions: Biological: OPT-822/OPT-821

INTERVENTIONS:
Biological: OPT-822/OPT-821

SUMMARY:
The purpose of this study is to evaluate the effect of OPT-822/OPT-821 on improving Progression-Free Survival (PFS) in subjects who have non-progressive epithelial ovarian, fallopian tube, or primary peritoneal cancer after cytoreductive surgery and platinum-based chemotherapy as initial treatment for primary disease or as salvage treatment for first relapse.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects ≥ 21 years of age with histologically confirmed ≥ stage II epithelial ovarian, fallopian tube, and primary peritoneal cancer at diagnosis
* Who have not progressed after initial treatment with cytoreductive surgery and at least 4 cycles of platinum-based chemotherapy.

OR

* Female subjects ≥ 21 years of age with first relapsed epithelial ovarian, fallopian tube, and primary peritoneal cancer (regardless of stage at diagnosis)
* Who have not progressed after received at least 4 additional cycles of platinum-based chemotherapy with or without having undergone secondary cytoreductive surgery .

Exclusion Criteria:

* Subjects with evidence of disease progression according to the GCIG CA125 criteria or RECIST 1.1 criteria.
* Subjects who are currently receiving any other concomitant anticancer therapy.
* Subjects with evidence of extra-abdominal metastasis.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Until disease progression or up to 5 years after the enrollment

SECONDARY OUTCOMES:
Disease Recurrence Rate | At 2 years after the enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan